CLINICAL TRIAL: NCT01211132
Title: Prospective Randomized Controlled Study of Cap Assisted Colonoscopy for the Detection of Colon Polyps
Brief Title: Cap Assisted Colonoscopy for the Detection of Colon Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Society for Gastrointestinal Endoscopy (Other)
Collaborators: Midwest Biomedical Research Foundation (Other)
Responsible Party: Amit Rastogi, MD (Prinicipal Investigator), Kansas City VA Medical Center
Organization: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AR0006
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Adenoma; Colon Polyps; Colon Cancer
Keywords: Colon polyps; Adenoma detection; Cap; Standard; Colon Cancer
MeSH Terms: conditions — Adenoma; Colonic Polyps; Colonic Neoplasms; Anterior polar cataract 2 | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cap arm (Active Comparator)
  Interventions: Device: Cap - Transparent retractable extension device.
- Standard arm (Active Comparator)
  Interventions: Device: Standard

INTERVENTIONS:
Device: Cap - Transparent retractable extension device. — Attaching a Cap - Transparent retractable extension device.
  Other Names: Cap Assisted Colonoscopy
  Arms: Cap arm
Device: Standard — Without attaching a transparent cap to the tip of colonoscope.
  Other Names: Standard Colonoscopy
  Arms: Standard arm

SUMMARY:
This simple technique of attaching a transparent cap to the tip of the colonoscope has been evaluated in Japan for improving the detection of polyps and cecal intubation but has not been formally evaluated in the US and other western countries. In one study (19), the polyp detection rate was higher with the transparent cap compared to no cap (49% vs. 39%, p=0.04). Also, the cecal intubation time was shorter with the cap (11.5 min vs 14 min, p=0.008). In a recently published study, a variation of the cap called the transparent retractable extension device was used (21). Overall, the number of adenomas detected were significantly higher with the device compared to without it (205 vs. 150, p=0.04). In an earlier study by Tada et al (22), use of a transparent cap improved the detection rate of lesions per patient (0.86 vs. 0.58) but did not increase the cecal intubation time. Finally, Lee et al (20) used cap assisted colonoscopy in patients with difficult colonoscopy procedure (defined as failure to pass through sigmoid colon after 20 minutes or failure to reach cecum). Using the cap, cecal intubation was achieved in 94% of patients and this proved to be an effective rescue method for failed or difficult colonoscopy. The major appeal of this technique is that it is inexpensive, very practical, and easy to use. Furthermore it is safe and there are no reported complications from this. If found to be effective in increasing the polyp yield it has the potential to being incorporated by busy gastroenterologists in their day to day clinical practice. These features and the preliminary data from Japan merit the evaluation of this promising technique in the US.

DETAILED DESCRIPTION:
The investigators hypothesize that adenoma detection rate will be higher using cap assisted colonoscopy compared to standard colonoscopy. Also, cap assisted colonoscopy will be safe and cecal intubation rate will be similar compared to standard colonoscopy.

Specific Aim 1 - To compare the prevalence of adenomas detected by standard colonoscopy and cap assisted colonoscopy.

Specific Aim 2 - To compare the number of adenomas detected per subject by standard colonoscopy and cap assisted colonoscopy.

Specific aim 3 - To compare the cecal intubation rate, insertion time, withdrawal time and complications of standard colonoscopy and cap assisted colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Referral for screening and/or surveillance colonoscopy and the ability to provide informed consent.

Exclusion Criteria:

* prior surgical resection of any portion of colon,
* prior history of colon cancer,
* history of inflammatory bowel disease,
* use of anti-platelet agents or anticoagulants that precludes removal of polyps during the procedure,
* poor general condition or any other reason to avoid prolonged procedure time
* inability to give informed consent,
* inadequate bowel preparation.
* history of polyposis syndrome or HNPCC,

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the prevalence of adenomas in the two groups. | 2 years

SECONDARY OUTCOMES:
The secondary outcomes are the number of adenomas detected per subject, cecal intubation rate, insertion times, withdrawal times and complication rates in the two arms. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Rastogi, MD, Principal Investigator — Veterans Affairs Medical Center, Kansas City, MO
Locations (1):
- Veterans Affairs Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Rastogi A, Bansal A, Rao DS, Gupta N, Wani SB, Shipe T, Gaddam S, Singh V, Sharma P. Higher adenoma detection rates with cap-assisted colonoscopy: a randomised controlled trial. Gut. 2012 Mar;61(3):402-8. doi: 10.1136/gutjnl-2011-300187. Epub 2011 Oct 13. PMID 21997547